CLINICAL TRIAL: NCT03454932
Title: Laboratory Research Study of the Immunosuppressive Effect of a Cell Therapy Product on PBMC Isolated From Blood of Patients With Inflammatory Rheumatic Diseases
Brief Title: Research Study on the Immunosuppressive Effects of a Cell Therapy Product on PBMC Isolated From Blood of Patients With Inflammatory Rheumatic Diseases
Status: Terminated | Type: Observational
Why Stopped: limited number of recruited patients
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: RAPSASPA-HBM
Record Dates: First submitted 2015-06-03; First posted 2018-03-06 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Spondylarthritis
Keywords: Rheumatoid Arthritis; Psoriatic Arthritis; Spondylarthritis; Rheumatic diseases; Inflammation; Autoimmune diseases; Osteoimmunology
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis; Rheumatic Diseases; Inflammation; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Rheumatoid Arthritis: Patients with Rheumatoid Arthritis
  Interventions: Other: Blood sampling
- Psoriatic Arthritis: Patients with Psoriatic Arthritis
  Interventions: Other: Blood sampling
- Spondylarthritis: Patients with Spondylarthritis
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling

SUMMARY:
Rheumatic diseases regroup a variety of disorders affecting the locomotor system including joints, muscles, connective tissues and soft tissues around the joints and bones. Inflammation and/or autoimmune reactions contribute to the aetiology of many rheumatic diseases. Such autoimmune conditions, commonly referred to as inflammatory rheumatic diseases (IRD), include arthritis of various origins such as rheumatoid arthritis (RA), psoriatic arthritis (PsA) or spondylarthritis (SpA). Patients with autoimmune diseases such as RA or SpA are in higher risk of fractures compared to the general population.

Initial pharmacotherapies for IRD remain NSAID treatment for pain relief, and anti-resorptive agents (e.g., TNF-alpha blockers) which aim at reducing bone loss and preventing occurrence of new bone erosions. Yet current treatments may have strong side effects and are not always effective (e.g., 35-40% of the patients treated with TNF-alpha inhibitors will initially or progressively loose response). Therefore there is a need for further treatment modalities in IRD, which would focus on both suppressing inflammation and treating bone disorders.

Current research studies indicate that Bone Therapeutics' allogeneic osteoblastic cells exhibit in vitro potent immunosuppressive and anti-inflammatory properties (in addition to osteo-regenerative and immune-privileged properties).

The present research study aims at investigating in vitro the properties of these osteoblastic cells in the context of inflammatory rheumatic diseases. In this purpose, in vitro assays will be used to test these immunosuppressive effects on peripheral blood mononuclear cells (PBMCs) of subjects diagnosed with RA, PsA and SpA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 18 years of age or older
* Subjects must belong to one of this group: Rheumatoid Arthritis (RA) Subjects OR Psoriatic Arthritis (PsA) Subjects OR Spondylarthritis (SpA) Subjects

Exclusion Criteria:

* Subjects diagnosed with other autoimmune/inflammatory diseases other than Crohn's disease, psoriasis, uveitis, Sjögren's syndrome and auto-immune thyroiditis
* Subjects with an active cancer and currently receiving a cancer treatment
* Women with known pregnancy
* Breastfeeding women
* Subjects with a known history of HIV and/or Hepatitis B and/or Hepatitis C infection and/or positive for HBs antigens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis, Psoriatic Arthritis and Spondylarthritis Subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04 (Actual); Study Completion 2017-06-04 (Actual)

PRIMARY OUTCOMES:
PBMC proliferation, as assessed with PBMC assay | 7 days
  Freshly prepared cell therapy product and PBMC will be mixed together in wells. Mixes will be incubated for 7 days in a humidified atmosphere of 5% CO2 in air at 37°C. PBMC proliferation will be assessed using tritiated (³H)-thymidine uptake (β-counter).
Secretion of pro-inflammatory cytokines (e.g., IL-1β) and anti- inflammatory cytokines (e.g., IL-10), as assessed with PBMC assay | 7 days
  Freshly prepared cell therapy product and PBMC will be mixed together in wells. Mixes will be incubated for 7 days in a humidified atmosphere of 5% CO2 in air at 37°C. Pro-inflammatory cytokines (e.g., IL-1β) and anti- inflammatory cytokines (e.g., IL-10) will be measured in culture supernatant using Luminex method.

SECONDARY OUTCOMES:
Record of past and current relevant medical history through questionnaire | time of first visit
Record of concomitant medications through questionnaire | time of first visit
Record of disease activity assessment (DAS28 and/or CASPAR and/or ASDAS and/or NY) | time of first visit
Record of any adverse events (if any) | time of first visit
  occurring during and/or after the blood sample collection procedure
Results of the laboratory blood tests for CBC, RF, CRP, HLA-B27 | 7 days
  Complete Blood Count (CBC), formula and electrolytes; Rheumatoid Factor (RF); C-Reactive Protein (CRP); HLA-B27